CLINICAL TRIAL: NCT06933459
Title: An Open Label, Randomized, Single Dose, 2-sequence, 2-period, Cross-over Phase 1 Study to Evaluate the Safety and Pharmacokinetics of AJU-C714 Compared to C714R in Healthy Adult Volunteers
Brief Title: To Evaluate the Safety and Pharmacokinetic Characteristics of AJU-C714 and C714R in Healthy Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AJU Pharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24PHL10102
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Drug Evaluation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Period 1: Reference Drug, single dose Period 2: Test Drug, single dose
  Interventions: Drug: Test Drug; Drug: Reference Drug
- Sequence B (Experimental): Period 1: Test Drug, single dose Period 2: Reference Drug, single dose
  Interventions: Drug: Test Drug; Drug: Reference Drug

INTERVENTIONS:
Drug: Test Drug — AJU-C714
Drug: Reference Drug — C714R

SUMMARY:
To evaluate the safety and pharmacokinetic characteristics of AJU-C714 and C714R in healthy adults

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult over 19 years of age and under 65 years of age.
2. Weight ≥ 50 kg (man) or 45 kg (woman), with calculated body mass index (BMI) of 18 to 30 kg/m2.
3. Those who have no congenital chronic disease or chronic disease requiring treatment and who have no pathological symptoms or findings.
4. Those who are eligible for clinical trials based on laboratory (hematology, blood chemistry, serum, urine test) and 12-lead ECG results during screening tests.
5. Those who voluntarily decide to participate and agree to comply with the cautions after hearing and fully understanding the detailed description of this clinical trial.
6. Those who agree to contraception during the participation of clinical trial.

Exclusion Criteria:

1. Those who take barbiturate and related (causing induction or inhibition of metabolism) drug within 1 month or the first administration of clinical trial drug within 10 days.
2. Those who received investigational product or bioequivalence test drug within 6 months before the first administration of clinical trial drug.
3. Those who donated whole blood within 8 weeks, received apheresis within 2 weeks, blood transfusion within 1 month or can't refrain from donating blood from the time of written consent until the end of the study.
4. Those who has a history of gastrointestinal disease or surgery which may affect the absorption of the drug.
5. Those who exceeding an alcohol consumption criteria Alcohol: Men - 21 glass/week, Women - 14 glass/week (1 glass: Soju 50 mL, Beer 250mL or liquor: 30mL), Smoke: 20 cigarettes/day.
6. Those who has under

   * Those who are hypersensitive to component of the Investigational product and have the medical history
   * Those with active liver disease or persistent elevation of aminotransferase levels of unknown
   * Those with myopathy
   * Those taking cyclosporin
   * Those with renal impairment with severe renal failure
   * Those with Hypothyroidism
   * Those who has Genetic problems such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption
7. Those who has a history of mental illness.
8. Those who are deemed unfit by the investigators to participate in the clinical trial for other reasons.
9. Women who are pregnant or who may be pregnant and breastfeed.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-05-24 (Actual); Primary Completion 2025-06-11 (Estimated); Study Completion 2025-06-24 (Estimated)

PRIMARY OUTCOMES:
AUCt of AJU-C714 | Pre-dose(0 hours), 3, 5, 10, 15, 20, 30, 40, 50 minutes, 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72 hours
Cmax of AJU-C714 | Pre-dose(0 hours), 3, 5, 10, 15, 20, 30, 40, 50 minutes, 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- H+ Yangji Hospital, Seoul, Republic of South Korea, Seoul, South Korea